CLINICAL TRIAL: NCT01241695
Title: Safety, Acceptability and Efficacy of a Long-term Intervention With a Diabetes-specific Low-carbohydrate, High-mono-unsaturated Fatty Acid Containing Oral Nutritional Supplement on Glycaemic Control in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GCOS-002-CFS
Record Dates: First submitted 2010-11-10; First posted 2010-11-16 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2010-11

CONDITIONS: Diabetes
Keywords: Oral nutritional supplement, diabetes mellitus type 2, glycaemic control; Oral nutritional supplement (Food for special medical purposes)
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Dietary Supplements; Food

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Diben DRINK (200 ml) / a diabetes-specific oral nutritional supplement
  Interventions: Dietary Supplement: Oral nutritional supplement, food for special medical purposes
- Control (Placebo Comparator): Fresubin(R) energy fibre DRINK / an isoenergetic standard oral nutritional supplement
  Interventions: Dietary Supplement: Oral nutritional supplement, food for special medical purposes

INTERVENTIONS:
Dietary Supplement: Oral nutritional supplement, food for special medical purposes — 2 servings of 200 ml per day, treatment period: 12 weeks
  Arms: Test
Dietary Supplement: Oral nutritional supplement, food for special medical purposes — 2 servings of 200 ml per day, treatment period: 12 weeks
  Arms: Control

SUMMARY:
The purpose of the study is to determine the safety, acceptability and the efficacy of a 12-week intervention with a diabetes-specific oral nutritional supplement on glycaemic control in type 2 diabetic patients with or at risk of malnutrition

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 2 diabetes according to the WHO diagnostic criteria for more than 6 months: Fasting plasma glucose (FPG) ≥ 126 mg/dl (7.0 mmol/l) or 2-h plasma glucose ≥ 200 mg/dl (11.1 mmol/l) during an OGTT (oral glucose tolerance test);
* HbA1c between 6.5-8.5 % (confirmed in the previous 3 months),
* capable of using oral nutritional supplementation,
* on stable and controlled anti-diabetic regime for at least 1 months,
* use of metformin and/or sulphonylureas as oral anti-diabetic medication,
* in need of nutritional support because of ≥5% involuntary weight loss in the last 3 months, ≥10% involuntary weight loss in the last 6 months, inadequate nutritional intake causing failure to meet nutritional requirements or at risk of developing malnutrition

Exclusion Criteria:

* diabetes type 1,
* participation in a clinical trial with an investigational product or regular use of disease-specific oral nutritional supplements within 4 weeks prior to study start
* patients requiring a fibre free diet,
* enteral tube feed or parenteral nutrition,
* concomitant therapy with systemic glucocorticoids, insulins or anti-diabetic medication other than metformin and sulphonylureas,
* known or suspected intolerance or allergy to any component of the investigational product(s),
* any acute gastrointestinal disease within 2 weeks prior to study entry,
* gastrectomy, gastroparesis or other gastric emptying abnormalities,
* acute sever heart failure (NYHA class 4), liver insufficiency / failure (male: ALAT > 150 U/l; female: ALAT > 120 U/l) or renal failure requiring dialysis,
* cancer cachexia,
* galactosaemia, fructosaemia,
* suspicion of drug abuse, abuse of/addiction to alcohol,
* pregnant or breast feeding women, or fertile women refusing to use contraceptives,
* patients with untreated major psychiatric disorder,
* known HIV positive (safety reasons),
* patient unable to co-operate adequately

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
postprandial blood glucose (iAUC) (0-240 min) | day 1
postprandial blood glucose (iAUC) (0-240 min) | day 42
postprandial blood glucose (iAUC) (0-240 min) | day 84

SECONDARY OUTCOMES:
postprandial peak blood glucose (0-240 min) | day 1, day 42, day 84
postprandial triglycerides (0-240 min) | day 1, day 42, day 84
total cholesterol, HDL-cholesterol, LDL-cholesterol | day 1, day 42, day 84
total protein, albumin, prealbumin | day 1, day 42, day 84
HbA1c, HOMA-IR index | day 1, day 42, day 84
c-peptide | day 1, day 84
gastrointestinal tolerance | week 1, week 6, week 12
palatability / taste test | week 1, week 6, week 12
  by means of a sensorial questionnaire the patients will evaluate the overall liking, appearance, smell, taste, mouth feel et cetera of the study nutrition.
daily compliance | day 1-84
  in a daily compliance questionnaire the patients record the amount of oral nutritional supplements consumed.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Mayr, Dr., Principal Investigator — Medical Practice, 78333 Stockach
Locations (1):
- Medical Practice, Stockach, Baden-Wurttemberg, Germany